CLINICAL TRIAL: NCT06836271
Title: The Effect of Cleaning the Biopsy Needle With Isopropyl Alcohol, Povidone Iodine and Formalin Before Transrectal Ultrasonography-guided Prostate Biopsy on Procedure-related Infective Complications
Brief Title: Cleaning the Biopsy Needle in TRUS Bx
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Mustafa Serdar CAGLAYAN, Assistant Professor Doctor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HititUrology001
Record Dates: First submitted 2025-01-30; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Prostatic Cancer
Keywords: Prostatic Neoplasms; Needle washing; Prostate biopsy; Sepsis
MeSH Terms: conditions — Prostatic Neoplasms; Sepsis | interventions — 2-Propanol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: 4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- biopsy needle with formalin (Experimental)
  Interventions: Combination Product: formaldehit
- biopsy needle with povidone iodine (Experimental)
  Interventions: Drug: Povidine-iodine
- Standart biyopsy (Active Comparator): No disinfection method is used in routine use in repetitive procedures when taking a transrectal biopsy.
  Interventions: Procedure: Standard BP control
- biopsy needle with isopropyl alcohol (Experimental)
  Interventions: Drug: Isopropyl Alcohol

INTERVENTIONS:
Drug: Isopropyl Alcohol — During repeated procedures while transrectal biopsy was being taken, the biopsy needle was disinfected with 70% Isopropyl alcohol every time it came into contact with the rectal mucosa.
  Arms: biopsy needle with isopropyl alcohol
Drug: Povidine-iodine — During repeated procedures while transrectal biopsy was being taken, the biopsy needle was disinfected with povidine-iodine every time it came into contact with the rectal mucosa.
  Arms: biopsy needle with povidone iodine
Combination Product: formaldehit — During repeated procedures while transrectal biopsy was being taken, the biopsy needle was disinfected with 10% formaldehit every time it came into contact with the rectal mucosa.
  Arms: biopsy needle with formalin
Procedure: Standard BP control — No disinfection method is used in routine use in repetitive procedures when taking a transrectal biopsy.
  Arms: Standart biyopsy

SUMMARY:
Prostate cancer(PCa) is the second most common cancer diagnosed in men. Clinical suspicion of PCa is mentioned in patients with digital rectal examination findings and elevated serum PSA. Despite all the advances in radiological imaging methods, the gold standard method in the diagnosis of the disease is systematic prostate biopsy performed under the guidance of transrectal ultrasonography, which is an invasive procedure.

In TRUS-guided transrectal prostate biopsy, bacteriuria may develop as a result of the rectum flora being injected into the urinary system through a biopsy needle. Infective complications may be encountered as a result of this contamination. Infective complications can present with conditions ranging from asymptomatic bacteriuria to sepsis.

A study has shown that disinfection of the biopsy needle with isopropyl alcohol reduces sepsis due to prostate biopsy compared to the standard procedure. In another study, disinfection of the biopsy needle tip with formalin was found to be associated with a decrease in infectious complications after transrectal prostate biopsy.

In this study, investigators aimed to conduct a prospective study comparing Transrectal Ultrasonography-guided Prostate Biopsy cases, in which the biopsy needle was cleaned with isopropyl alcohol, povidone iodine and formalin, and standard biopsy patients in terms of infectious complications.

DETAILED DESCRIPTION:
Objective To reduce procedure-related infective complications after Transrectal Ultrasonography-guided Prostate Biopsy Method Prostate cancer is the second most common cancer diagnosed in men. In 2020, approximately 1.4 million people were diagnosed worldwide [1,2]. The number of PCa detected by autopsy is roughly the same worldwide [3]. In a systematic review of autopsy studies, the prevalence of PCa under the age of 30 years was reported to be 5% (confidence interval-CI: 95%), with a 1.7 (1.6-1.8) (odds ratio-OR) fold increase per 10 years, reaching 59% (48-71%) over the age of 79 years [4].

Clinical suspicion of PCa is mentioned in patients with finger rectal examination findings and elevated serum PSA. Despite all the advances in radiologic imaging modalities, the gold standard method for the diagnosis of the disease is systematic prostate biopsy under transrectal ultrasonography guidance, which is an invasive procedure. [5]

Transrectal ultrasonography (TRUS) was first described by Wild and Reid in 1957. TRUS plays an important role in prostate diseases as it is inexpensive, easily applicable and guides biopsy. Conventional TRUS-guided prostate biopsy is performed with 12 pieces of tru-cut samples taken systematically and randomized.

Although it can be safely performed in the outpatient setting and is easily tolerated by patients, Transrectal Ultrasonography-guided Prostate Biopsy can lead to serious complications such as hematuria, rectal bleeding, acute urinary retention, urinary tract infection and sepsis.

Urinary tract infection accompanied by fever is the most common complication after biopsy. Bacteriuria after prostate biopsy is reported between 20% and 50% in the literature. [6] Several studies have shown that antibiotic prophylaxis largely prevents infection. [6,7]

During TRUS-guided transrectal prostate biopsy, bacteriuria may develop as a result of the rectal flora being introduced into the urinary system through the biopsy needle. Infective complications may occur as a result of this transmission. Infective complications can range from asymptomatic bacteriuria to sepsis.

In one study, disinfection of the biopsy needle with isopropyl alcohol was shown to reduce prostate biopsy-related sepsis compared to the standard procedure. [8] In another study, disinfection of the biopsy needle tip with formalin was associated with a decrease in infectious complications after transrectal prostate biopsy.[9] In this study, investigators aimed to prospectively examine the infectious complications occurring in a total of 200 cases of Transrectal Ultrasonography-guided Prostate Biopsy to be performed in our clinic in 2025.

In 200 patients who underwent Trans Rectal Ultrasonography-guided prostate biopsy procedure, infective parameters, signs and symptoms such as fever, dysuria, and possible complications such as hospitalization requirement, sepsis will be prospectively investigated to evaluate postop infective complications of disinfection of the biopsy needle with formalin, povidone iodine or isopropyl alcohol before each biopsy.

In the study, each patient will undergo bt-enema for bowel cleansing before the procedure, rectal cleansing with povidone iodine, and prophylactic antibiotherapy will be started 3 days before the procedure. Patients will be randomly divided into four groups, 50 patients will be disinfected with Bx needle formalin before the procedure, 50 patients will be disinfected with Bx needle povidone iodine before the procedure, 50 patients will be disinfected with Bx needle isopropyl alcohol before the procedure, and the other 50 patients will not be disinfected with isopropyl alcohol, povidone iodine or formalin as in the standard practice. In the first 1 week after the procedure, their symptoms will be questioned by daily phone calls. Within 1 week, complete urinalysis and urine culture will be obtained from symptomatic patients (burning during urination, fever, chills, chills). Patients with a fever above 37.8 will be hospitalized after a complete urine test, urine and blood culture. On day 14, outpatients will be called for outpatient follow-up and patients without any symptoms will be lost to follow-up.

Estimated completion time of the study 6 months Inclusion criteria

* Oriented-coopere patients
* Patients without active urinary tract infection - Patients without active urinary tract infection
* Patients without bleeding diathesis
* Patients who accept the study Exclusion criteria
* Patients with active urinary tract infection
* Patients with bleeding diathesis
* Patients with sonal or cystofix
* Patients with a history of previous prostate surgery Determination of sample size For the main (Primary) hypothesis in our study (The effect of cleaning the biopsy needle with isopropyl alcohol, formalin and povidone iodine before Transrectal Ultrasonography-guided Prostate Biopsy on procedure-related infective complications), power analysis was performed using f-test in independent groups. In order to reach 95% power with α=0.05 error (two-way hypothesis), it was determined that a minimum total of 176 patients were needed as a result of the power analysis calculated using Cohen's d=0.25 effect size calculated by using the literature information. In this study, investigators decided to enroll a total of 200 patients, with a minimum of 50 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Oriented-coopere patients
* Patients without active urinary tract infection - Patients without active urinary tract infection
* Patients without bleeding diathesis
* Patients who accept the study

Exclusion Criteria:

* Patients with active urinary tract infection

  * Patients with bleeding diathesis
  * Patients with sonal or cystofix
  * Patients with a history of previous prostate surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Determination of sample size | 6 months
  For the main (Primary) hypothesis in our study (The effect of cleaning the biopsy needle with isopropyl alcohol, formalin and povidone iodine before Transrectal Ultrasonography-guided Prostate Biopsy on procedure-related infective complications), power analysis was performed using f-test in independent groups. In order to reach 95% power with α=0.05 error (two-way hypothesis), it was determined that a minimum total of 176 patients were needed as a result of the power analysis calculated using Cohen's d=0.25 effect size calculated by using the literature information. In this study, we decided to enroll a total of 200 patients, with a minimum of 50 in each group. Patients will be evaluated with a post-operative survey. Patients will be followed for 4 weeks after the operation.